CLINICAL TRIAL: NCT03410628
Title: Non-invasive Neurostimulation of the Vagus Nerve With the gammaCore Device for the Relief of Pain and Allodynia Associated With Migraine
Brief Title: Non-invasive Neurostimulation for the Relief of Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-SA-01
Record Dates: First submitted 2015-03-12; First posted 2018-01-25 (Actual); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gammaCore Active Device (Experimental): open label
  Interventions: Device: gammaCore

INTERVENTIONS:
Device: gammaCore — Non-invasive vagal nerve stimulator

SUMMARY:
The purpose of this feasibility study is to gather preliminary information on the safety and effectiveness of patient self-administration of a noninvasive neurostimulation of the vagus nerve using the GammaCore device for the treatment of pain and allodynia symptoms associated with acute migraine in adults.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, unblinded, multi-center feasibility study; 25 subjects will be enrolled at up to 5 study centers. Subjects considered for participation in this study will be those who have a diagnosis and documented history at least 2 episodes of acute headache pain and allodynia associated with migraine per month, but no more than 15 headache days per month. Subjects may, but are not required to experience prodromal symptoms, such as aura, or concomitant photophobia, phonophobia, or nausea with their migraine episodes, so long as their headaches meet the IHS-Classification criteria for migraine. Subjects will be screened for study eligibility and consented for study participation at presentation to the headache clinic. Once consented, subjects will be trained by the Investigator(s) at the study center on at-home use of the GammaCore device and on study data collection and other requirements.

Each subject enrolled in this study will treat up to 3 migraine headaches at home over a period of up to 6 weeks.

From the onset of headache pain, the subject will withhold usual migraine medications and wait until the pain becomes moderate or severe, or 30 minutes, whichever is sooner. At that point, the subject will self-administer a first stimulation treatment, which is 90 seconds in duration.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 55 years.
* Has been previously diagnosed as suffering from migraine, in accordance with the IHS-Classification criteria (2nd) (with or without aura).
* Experiences at least 2 migraines per month, but less than 15 headache days per month (over the last 3 months).
* Has age of onset of migraine less than 50 years old.
* Is able to distinguish migraines from other headaches (e.g. tension headache).
* Agrees to withhold usual migraine medications until after stimulation treatment with the GammaCore device.
* Agrees to follow all of the requirements of the study, including follow-up visit requirements, and is sufficiently trained with respect to the operation of the GammaCore device and the data collection procedures.
* Agrees to report use of the GammaCore device, study data, and any adverse device effects to the study center within 24 hours of treatment(s), and agrees to schedule an office visit 4-10 days after the third and final treatment, or when 6 weeks has passed, whichever comes first.
* Is able to give written Informed Consent, or his/her legally authorized representative is available to give written Informed Consent.

Exclusion Criteria:

* Has a history of aneurysm, bleed, brain tumors or significant head trauma.
* Has a lesion (including lymphadenopathy) at the therapy head placement site.
* Has known or suspected severe atherosclerotic cardiovascular disease, carotid artery disease (e.g. bruits or history of TIA or CVA) or congestive heart failure (CHF).
* Has a history of epilepsy.
* Has suspected or confirmed sepsis, or infection.
* Has a clinically significant irregular heart rate or rhythm.
* Is receiving pressors to maintain blood pressure.
* Has a history of syncope.
* Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Has been implanted with metal cervical spine hardware.
* Has a history of carotid endarterectomy or vascular neck surgery on the right side.
* Has a condition that would interfere with headache pain self-assessment.
* Is pregnant or is thinking of becoming pregnant in the next 6 weeks.
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
* Takes medication for acute headaches more than 10 days per month.
* Has a history or suspicion of substance abuse
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | gammaCore Active Device
Started | 21
Completed | 15
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | gammaCore Active Device
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 38.6 [22 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17
  Asian | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 21

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Adverse Events
Description: Safety was assessed by collecting adverse events for the duration of the study
Time Frame: Up to 4 months
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore Active Device
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Change in Headache Pain Severity From Baseline to 120 Minutes for First Treated Migraine Attack
Description: At the onset of headache pain subjects self-administered treatment with the study device and completed headache pain scores using a 4 point scale (where 3 = severe, 2 = moderate, 1 = mild and 0 = no pain) at baseline (0 minutes) and 120 minutes.
Time Frame: 120 minutes
Population: Safety population, 6 subjects had missing data
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | gammaCore Active Device
Number analyzed (Participants) | 15
units on a scale
  Headache pain severity at Baseline | 2.2 [1 to 3]
  Headache pain severity at 120 minutes | 1.2 [0 to 3]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | gammaCore Active Device
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore Active Device (N=21)
Diarrhea (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less